CLINICAL TRIAL: NCT02453620
Title: A Phase 1 Study Evaluating Safety, Tolerability, and Preliminary Antitumor Activity of Entinostat and Nivolumab With or Without Ipilimumab in Advanced Solid Tumors
Brief Title: Entinostat, Nivolumab, and Ipilimumab in Treating Patients With Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery or Locally Advanced or Metastatic HER2-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00741; NCI-2015-00741 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SKCCC J15221; L9844; J15221; 9844 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 9844 (Other: CTEP); UM1CA186689 (NIH); UM1CA186690 (NIH); UM1CA186691 (NIH); UM1CA186717 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Breast Adenocarcinoma; Invasive Breast Carcinoma; Malignant Solid Neoplasm
MeSH Terms: interventions — Biopsy; Blood Specimen Collection; entinostat; Ipilimumab; CTLA-4 Antigen; Nivolumab; Pharmacogenomic Testing; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (entinostat, nivolumab, ipilimumab) (Experimental): Patients receive entinostat PO on days -14 and -7 and then weekly, nivolumab IV over 60 minutes on day 1 and then every 2 weeks, and ipilimumab IV over 90 minutes on day 1 and then every 6 weeks for 4 doses. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT as clinically indicated throughout the trial. Patients may undergo PET/CT or bone scan throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Other: Blood Sample; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Entinostat; Biological: Ipilimumab; Biological: Nivolumab; Other: Pharmacogenomic Study; Other: Pharmacological Study; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Other: Blood Sample — Undergo blood sample collection
  Other Names: Blood; Blood Draw; Blood Specimen
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS 275; MS-275; MS275; SNDX 275; SNDX-275; SNDX275
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Other: Pharmacological Study — Correlative studies
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial studies the side effects and best dose of entinostat and nivolumab when given together with ipilimumab in treating patients with solid tumors that have spread to other places in the body and usually cannot be cured or controlled with treatment (metastatic) or that cannot be removed by surgery (unresectable) or human epidermal growth factor receptor 2 (HER2)-negative breast cancer that has spread from where it started to nearby tissue or lymph nodes or other parts of the body. Entinostat is in a class of drugs called histone deacetylase (HDAC) inhibitors. It may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth (locally advanced/metastatic). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving entinostat and nivolumab together with ipilimumab may work better in treating in patients with solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination of entinostat and nivolumab with or without ipilimumab in subjects with advanced solid tumors.

II. To determine the recommended phase II dose (RP2D) of the combination of entinostat and nivolumab with ipilimumab in subjects with advanced solid tumors and to further confirm the safety of the combination therapy in subjects with advanced HER2-negative breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate whether treatment with entinostat alone or in combination with nivolumab and ipilimumab results in an increase in the ratio of tumor antigen-specific effector T cells (Teff) to regulatory T cell (Treg) in tumor biopsies compared to baseline.

II. To describe preliminary anti-tumor activity of entinostat and nivolumab in combination with or without ipilimumab in patients with advanced solid tumors.

III. To assess preliminary anti-tumor activity in an expansion cohort of patients with advanced breast cancer treated at the RP2D.

EXPLORATORY OBJECTIVES:

I. To explore changes in immune-related biomarkers (e.g., expression of checkpoint receptors [PD-1/PD-L1], the number of myeloid derived suppressor cells [MDSCs], inflammatory T cell signature, T cell receptor [TCR] repertoire) in tumor biopsies or peripheral blood lymphocytes (PBL) pre- and post-therapy.

II. To correlate changes in immune-related biomarkers pre- and post-combination therapy with response.

III. To measure tumor-specific mutations and mutant neo-antigens recognized by patient T cells in tumor biopsies and to describe association with response.

IV. To evaluate changes in frequency of T cells recognizing tumor-specific mutant neo-antigens in peripheral blood lymphocytes (PBL) pre- and post-therapy.

V. To evaluate changes in candidate gene expression, including the azacitidine (AZA) immune genes (AIM genes) in malignant tissue, gene methylation silencing in circulating deoxyribonucleic acid (DNA) and malignant tissue pre- and post-therapy.

VI. To correlate the pharmacodynamic outcomes (e.g., safety, efficacy, and changes in gene methylation status) with the exposure of entinostat (i.e., pharmacokinetics) when co-administered with nivolumab with or without ipilimumab.

VII. To conduct pharmacogenomic association analyses to assess the potential clinical utility of CD86 gene polymorphisms as genetic determinants of immune mediated adverse events.

OUTLINE: This is a dose-escalation study.

Patients receive entinostat orally (PO) on days -14 and -7 and then weekly, nivolumab intravenously (IV) over 60 minutes on day 1 and then every 2 weeks, and ipilimumab IV over 90 minutes on day 1 and then every 6 weeks for 4 doses. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) as clinically indicated throughout the trial. Patients may undergo positron emission tomography (PET)/CT or bone scan throughout the trial. Patients also undergo tissue biopsy and blood sample collection during screening and on the trial.

After completion of study treatment, patients are followed up every 3 months until disease progression and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation: patients must have histologically or cytologically confirmed solid tumor malignancy that is metastatic or unresectable and for whom either standard curative or palliative measures do not exist or are no longer effective, or for whom anti-PD-L1/cytotoxic T-lymphocyte antigen (CTLA)-4 is appropriate
* Dose expansion: patients must have histologically or cytologically confirmed invasive adenocarcinoma of the breast (human epidermal growth factor receptor 2 [HER2]-negative) that is locally advanced/metastatic and has progressed despite standard therapy; at least 1 prior chemotherapy regimen in the metastatic setting, and two lines of hormonal therapy (administered in the adjuvant or metastatic setting) for patients with hormone receptor-positive disease; NOTE: HER2-negativity will be defined per American Society of Clinical Oncology (ASCO)-College of American Pathologists (CAP) guidelines; patients whose tumors have HER2 immunohistochemistry (IHC) 3+, in situ hybridization (ISH) >= 2.0, or average HER2 copy number >= 6.0 signals per cell are not eligible
* Age ≥ 18 years.

  * NOTE: Because no dosing or adverse event data are currently available on the use of these agents in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Karnofsky >= 70%)
* Life expectancy of greater than 12 weeks
* Hemoglobin (HgB) >= 9.0 g/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN); an exception to this may be allowed for participants with Gilbert's syndrome with documented approval by the protocol chair
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min using the modified Cockcroft-Gault formula
* Negative (serum or urine) pregnancy test, for women of childbearing potential only
* Patients must have measurable or evaluable/non-measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; patients with bone only disease are not eligible due to difficulties in obtaining serial bone biopsies for correlative analyses; NOTE: for patients with metastatic disease in the liver, tumor burden should not be deemed significant (e.g., to no more than 30% of total liver volume as assessed by local review/investigator)
* Adequate pulmonary function as assessed by oxygen saturation >= 90% when ambulating and not requiring supplemental oxygen
* Patient must have an accessible non-bone tumor lesion from which serial core biopsy specimen can be obtained; NOTE: if baseline biopsy is attempted and is unsuccessful (e.g., patient intolerance, inadequate tissue), the patient will still be considered eligible for the study; if core biopsy is not possible, other methods may be approved in advance by the protocol chair/designee
* The effects of nivolumab, ipilimumab and entinostat on the developing human fetus are unknown; for this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at baseline; women must not be breastfeeding; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception; NOTE: A WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes
* Willingness to provide tissue and blood samples for mandatory translational research
* Willingness to return to the enrolling institution for follow-up
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or other systemic therapy or radiotherapy, or those who have not recovered from adverse events due to prior administered agents as follows:

  * Chemotherapy < 3 weeks prior to registration
  * Hormone therapy < 2 weeks prior to registration
  * Targeted therapy (other than below) < 2 weeks prior to registration (e.g., tyrosine kinase inhibitors)
  * Trastuzumab < 6 weeks prior to registration
  * Bevacizumab < 6 weeks prior to registration
  * Nitrosoureas/mitomycin C < 6 weeks prior to registration
  * Radiotherapy < 3 weeks prior to registration (NOTE: a previously irradiated lesion may not be used as a target lesion unless there is evidence of post-radiation progression)
  * Surgery < 3 weeks prior to registration
  * Other approved or investigational agents < 3 weeks prior to registration unless otherwise noted by the protocol chair
  * Patients who have received prior epigenetic (e.g., histone deacetylase [HDAC] inhibitors such as entinostat, panobinostat, vorinostat, romidepsin or demethylating agents such as 5-azacitidine or decitabine) immunomodulatory or other checkpoint inhibitors should only be considered after discussion with the protocol chair
  * Those who have not recovered from acute adverse events to grade < 2 or baseline due to agents administered, with exception of alopecia, unless approved by the protocol chair
* Known sensitivity to or history of allergic reactions attributed to compounds of similar chemical or biologic composition entinostat, nivolumab, or ipilimumab; history of severe hypersensitivity reaction to any monoclonal antibody
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis, systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, autoimmune hepatitis, and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* NOTE: patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity; NOTE: subjects must have baseline oxygen/saturation level requirements as above
* Patients with active or untreated brain metastases or leptomeningeal metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; NOTE: Patients with previously treated brain metastases must have stable neurologic status and magnetic resonance imaging (MRI) imaging following local therapy (surgery or radiation) for at least 4 weeks, with no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration (stable low dose dexamethasone allowed at discretion of protocol chair)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that in the judgment of the investigator would limit compliance with study requirements
* Pregnant women are excluded from this study because the agents have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued
* Known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; patients who have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C antibody (HCV Ab)/ribonucleic acid (RNA) (HCV RNA) indicating acute or chronic infection are also ineligible (baseline testing required); these are because of the potential for pharmacokinetic interactions with the study agents; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients requiring concurrent administration of valproic acid are also excluded
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study
* Another active malignancy =< 3 years prior to registration with the exception of non-melanotic skin cancer or carcinoma-in-situ of any type; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer; any malignancy considered to be indolent and that has never required therapy may allowed at the discretion of the protocol chair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events of entinostat and nivolumab in combination with ipilimumab | Up to 100 days after last dose of nivolumab
  Graded per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Safety and tolerability will be analyzed through the incidence of adverse events, serious adverse events, and specific laboratory abnormalities (worst grade) in each arm. Toxicities will be tabulated by type and grade for all doses and presented using frequencies and percentages based on the CTCAE v5.0. The proportion of dose-limiting toxicities at each dose level will be reported with exact 95% confidence intervals.

SECONDARY OUTCOMES:
Changes in ratio of effector T cell (Teff) to regulatory T cell (Treg) in tumor biopsies | Baseline to up to 2 weeks post-entinostat
  Measured by immunohistochemistry (IHC) staining of paraffin embedded tumor specimens. Changes will be treated as a continuous variable and summarized with descriptive statistics. Changes will also be graphically depicted using exploratory plots (e.g. bar plots, boxplots) and means will be estimated with 95% confidence intervals. A paired t-tests or nonparametric Wilcoxon signed-rank test may be used to determine whether or not the data shows evidence of changes from baseline.
Objective response rate | Up to 5 years
  Defined as the total number of patients with either complete response (CR) or partial response (PR) divided by the total number of patients in the population of interest (expansion cohort of patients with advanced breast cancer). Tumor assessment will be based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 and immune related response criteria (irRC).
Disease control rate (expansion cohort of patients with advanced breast cancer) | Up to 5 years
  Defined as the percentage of patients who have achieved CR, PR or stable disease (SD) among all response evaluable patients based on RECIST v1.1 and irRC. Estimated by the number of patients who achieve a confirmed response plus the number of patients who have stable disease for a duration of at least 6 months divided by the total number of evaluable patients.
Progression-free survival (PFS) | Time from start of treatment to time of disease progression or death, whichever occurs first, assessed at 6 months
  Defined as the proportion of patients remaining alive and free of disease progression (expansion cohort of patients with advanced breast cancer). Exact binomial 95% confidence intervals will be provided. The distribution of PFS, duration of response, and duration of stable disease will be described using the method of Kaplan-Meier, if warranted. Advanced breast cancer patients in the dose escalation portion treated at the recommended phase 2 dose (RP2D), if any, will be pooled with patients in the dose expansion cohort for these analyses.
Duration of overall response (expansion cohort of patients with advanced breast cancer) | Time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or death, assessed up to 5 years
  Duration of response will be described using the method of Kaplan-Meier, if warranted. Advanced breast cancer patients in the dose escalation portion treated at the RP2D, if any, will be pooled with patients in the dose expansion cohort for these analyses.
Duration of stable disease (expansion cohort of patients with advanced breast cancer) | Time measurement criteria are met for SD until the first date that recurrent or progressive disease is objectively documented or death, assessed up to 5 years
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 and immune related response criteria (irRC). Duration of stable disease will be described using the method of Kaplan-Meier, if warranted. Advanced breast cancer patients in the dose escalation portion treated at the RP2D, if any, will be pooled with patients in the dose expansion cohort for these analyses.

OTHER OUTCOMES:
Changes in number of myeloid derived suppressor cells (MDSCs) in peripheral blood and tumor biopsies | Baseline to up to 8 weeks
  Measured by flow cytometry pre and post-therapy. Summarized with descriptive statistics and graphically displayed by exploratory plots for overall and by tumor type if warranted. Changes will be estimated as a ratio change (post/pre) and data will be log transformed as appropriate. Difference between pre- and post-therapy will be explored using paired t-tests or Wilcoxon signed rank tests as appropriate for continuous variables and McNemar's test for dichotomous or categorical variables. Distributions of immune parameters across clinical responders and non-responders will be evaluated and graphically displayed using box plots.
Post-combination therapy expression of checkpoint inhibitors (PD-1/PD-L1) in tumor biopsies | Up to 8 weeks
  Measured by immunohistochemistry (IHC). Summarized with descriptive statistics and graphically displayed by exploratory plots for overall and by tumor type if warranted. Changes will be estimated as a ratio change (post/pre) and data will be log transformed as appropriate. Difference between pre- and post-therapy will be explored using paired t-tests or Wilcoxon signed rank tests as appropriate for continuous variables and McNemar's test for dichotomous or categorical variables. Distributions of immune parameters across clinical responders and non-responders will be evaluated and graphically displayed using box plots.
Changes in other immune-related biomarkers (e.g., ratio of effector T cells: regulatory T cells, inflammatory T cell signature, T cell receptor [TCR] repertoire) in tumor biopsies or peripheral blood lymphocytes (PBL) pre and post therapy | Baseline to up to 8 weeks
  Summarized with descriptive statistics and graphically displayed by exploratory plots for overall and by tumor type if warranted. Changes will be estimated as a ratio change (post/pre) and data will be log transformed as appropriate. Difference between pre- and post-therapy will be explored using paired t-tests or Wilcoxon signed rank tests as appropriate for continuous variables and McNemar's test for dichotomous or categorical variables. Distributions of immune parameters across clinical responders and non-responders will be evaluated and graphically displayed using box plots.
Tumor-specific mutations and mutant neo-antigens recognized by patient T cells in tumor biopsies | Up to 8 weeks
  Measured by whole-exome sequencing.
Changes in frequency of T cells recognizing tumor-specific mutant neo-antigens in tumor biopsies pre and post-therapy | Baseline to up to 8 weeks
Changes in candidate gene re-expression in malignant tissue, gene methylation silencing in circulating deoxyribonucleic acid (DNA) and malignant tissue pre and post-therapy | Baseline to up to 8 weeks
  Changes will be estimated as a ratio change (post/pre) and data will be log transformed as appropriate to induce symmetry and stabilize the variability. Difference between pre- and post-therapy will be explored using paired t-tests or Wilcoxon signed rank tests as appropriate for continuous variables and McNemar's test for dichotomous or categorical variables. Distributions of immune parameters across clinical responders and non-responders will be evaluated and graphically displayed using box plots. Change in these parameters with tumor response evaluated using Jonckheere-Terpstra trend test, Wilcoxon rank sum test as well as logistic regression where appropriate.
Pharmacodynamic outcomes (e.g., safety, efficacy, and changes in gene methylation status) with the exposure of entinostat when coadministered with nivolumab with or without ipilimumab | Up to 5 years
  Association of baseline and change in these parameters with clinical response will be evaluated using Wilcoxon rank sum tests.
CD86 gene polymorphisms as genetic determinants of immune mediated adverse events | Up to 8 weeks
  Pharmacogenomic association analyses will be performed using Fisher's exact test or Cochran-Armitage trend test to explore the potential clinical utility of CD86 gene polymorphisms as genetic determinants of immune mediated adverse events. Methods such as logistic or proportional hazards regression will likely be used for these analyses as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Roisin M Connolly, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania